CLINICAL TRIAL: NCT03384082
Title: A Randomised Controlled Trial of Hysteroscopic Resection of Mild Septum/Arcuate Uteri in Women With Recurrent Miscarriage.
Brief Title: A Randomised Controlled Trial of Hysteroscopic Resection of Mild Septum/Arcuate Uteri.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Song Dongmei, Principal Investigator, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FuXingH02
Record Dates: First submitted 2017-12-13; First posted 2017-12-27 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Arcuate Uterus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hysteroscopic treatment (Experimental): Hysteroscopic surgery
  Interventions: Procedure: hysteroscopic treatment
- Control group (No Intervention): No treatment

INTERVENTIONS:
Procedure: hysteroscopic treatment — treatment
  Arms: Hysteroscopic treatment

SUMMARY:
At least 82 cases of recurrent miscarriage women with a diagnosis of arcuate uterus, confirmed by three-dimensional intra-vaginal sonography (3D-TVS) and hysteroscopy, will be recruited. The subjects will be randomly divided into two groups, the experimental group will be given hysteroscopic treatment, the control group will receive no treatment. The pregnancy rates (>12 weeks) of the two groups will befollowed and compared.

DETAILED DESCRIPTION:
This study will be carried out at the Hysteroscopy center of the Fuxing Hospital, Beijing, China. At least 82 recurrent miscarriage women with a diagnosis of arcuate uterus who had unexplained recurrent spontaneous abortion (less than 12 weeks) before and have fertility requirement will be recruited. The patients will be explained the study and sign the informed consent. According to the random number table, the corresponding cases were divided into treatment group and control group. The experimental group will be given hysteroscopic treatment, the control group will receive no treatment. The follow up of the spontaneous abortion rate and the pregnancy rate of two groups will be screened within 1-2 years and the correlation between the arcuate uterus and recurrent miscarriage will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Women with arcuate/mild septum uteri
2. Women with unexplained recurrent miscarriage (less than 12 weeks)
3. Having a second time fertility requirement
4. Having Informed consent before entering this study, and be willing to receive hysteroscopic treatment

Exclusion Criteria:

1. 3D-TVS and hysteroscopy suggest uterine fibroids (submucosal and III type uterine fibroids, intramural fibroids,the diameter of whichis greater than 4cm), adenomyosis, endometrial polyps, intrauterine adhesions and other uterine factors that may lead to spontaneous abortion
2. Endometrial pathological diagnosis of chronic endometritis, endometrial hyperplasia and endometrial cancer
3. Ultrasound or HSG suggest hydrosalpinx
4. Chromosome abnormalities of the couples, positive findings of pre-thrombosis state and the detection of immunity, uterine malformation, uterine fibroids, adenomyosis and other uterine factors causing recurrent miscarriage
5. Semen abnormality in male
6. FSH > 10

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The pregnancy rate(>12 weeks)of the two groups | 2 years
  The pregnancy rate(>12 weeks) of the two groups after receiving hysteroscopic treatment and no treatment.
The spontaneous abortion rate of the two groups | 2 years
  The spontaneous abortion rate of the two groups after receiving hysteroscopic treatment and no treatment.
The live birth rate of the two groups | 2 years
  Te live birth rate of the two groups after receiving hysteroscopic treatment and no treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Song, Ph.D, Study Chair — Fuxing Hospital, Capital Medical University; Tinchiu Li, Ph.D, Study Director — Prince of Wales Hospital, Chinese University of Hong Kong
Locations (1):
- Hysteroscopic Centre of Fuxing Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP